CLINICAL TRIAL: NCT00899522
Title: Fanconi Anemia Cancer Cell Repository
Brief Title: Tissue Sample Collection From Patients With Fanconi Anemia
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Grover Bagby, Professor Emeritus, OHSU Knight Cancer Institute
Other Study IDs: IRB00001100; P30CA069533 (NIH); OHSU-HEM-03022-LX; OHSU-IRB00001100; OSHU-CR00003822; CDR0000445453 (Other: NCI PDQ)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-11

CONDITIONS: Fanconi Anemia; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: Fanconi anemia; unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Fanconi Anemia | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

INTERVENTIONS:
Other: biologic sample preservation procedure — Once the pathologist has taken the material needed to establish diagnosis of cancer, the anonymized snap-frozen and fresh samples will be either shipped to our laboratory for analysis or will be picked up by a member of the principal investigator's lab team. Samples will be stored indefinitely.
Procedure: biopsy — Once the pathologist has taken the material needed to establish diagnosis of cancer, 1-10 grams of the remaining tissue should be placed in phosphate buffered saline and shipped to the Bagby Lab.

SUMMARY:
RATIONALE: Collecting and storing samples of tumor tissue from patients with Fanconi anemia to test in the laboratory may help the study of cancer in the future.

PURPOSE: This laboratory study is collecting and storing tumor tissue samples from patients with Fanconi anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Acquire rare solid tumor samples from patients with Fanconi anemia in order to create a Fanconi Anemia Cell Repository at the Oregon Health and Science University Cancer Institute.
* Study repository tissue using a variety of molecular methods, including gene microarrays.
* Develop cancer cell lines that are publicly available from tissue archived from patients with Fanconi anemia.

OUTLINE: Tumor biopsies are collected from patients with Fanconi anemia and archived for future molecular studies, cell line generation, and general usage by the research community at large. Medical information about the patient's cancer is also archived.

PROJECTED ACCRUAL: Not specified.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed Fanconi anemia
* Confirmed malignant solid tumor
* Biopsy of tumor tissue available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 1 Year to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: To recruit participants into this project, an announcement will be posted on the Fanconi Anemia Research Fund website (http://www.fanconi.org/) after IRB approval is obtained.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2005-08; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Creation of a Fanconi Anemia Cell Repository using rare solid tumor samples from patients with Fanconi anemia | Duration of the study
Study tissue samples by molecular methods, including gene microarrays | Duration of the study
Development of cancer cell lines from tissue archived from patients with Fanconi anemia | Duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Grover C. Bagby, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon, United States